CLINICAL TRIAL: NCT00606814
Title: A Phase I Study of IPI-504 and Docetaxel in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of IPI-504 and Docetaxel in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-504-05; IPI-504-05
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Solid Tumors
Keywords: Solid Tumors, IPI-504, docetaxel,cancer
MeSH Terms: conditions — Neoplasms | interventions — tanespimycin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: IPI-504, docetaxel — 1. IPI-504 administered IV at a dose of 300mg/m2
  2. Docetaxel at a fixed dose of 75 mg/m2 for every 3 weeks dose administration or 36 mg/m2 for weekly administration
  Other Names: Taxotere

SUMMARY:
This study is a Phase I clinical trial of IPI-504 in combination with docetaxel (Taxotere).The purposes of the study are to determine:

* the safety profile,
* the highest dose of IPI-504 that can be given with docetaxel without causing severe side effects, and
* to recommend a Phase II dose of the combination in patients with solid tumors.

DETAILED DESCRIPTION:
IPI-504 is a novel small molecule inhibitor of heat shock protein 90 (Hsp90), an emerging and recently identified target for cancer therapy. Hsp90 is a protein chaperone that plays a central role in maintaining the proper folding, function and viability of various "client proteins". Many of the client proteins stabilized by Hsp90 are oncoproteins and cell-signaling proteins important in cancer cell proliferation and cancer cell survival.

This is a multi-center, open-label, dose escalating study in which patients will be treated with a fixed dose of docetaxel followed by IPI-504 following one of three dosing schedules.

Once an MTD has been defined, up to 20 additional patients with non-small cell lung cancer (NSCLC) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed malignancy that is metastatic or unresectable, for which one of the two statements must apply:

  * Standard therapy able to provide clinical benefit does not exist or is no longer effective AND / OR
  * Single agent docetaxel would be appropriate therapy.
* Progressive disease with development of new lesions or an increase in preexisting lesions on CT, MRI, PET, bone scintigraphy, or by physical examination.
* Measurable disease by RECIST criteria with the exception of prostate cancer patients.
* >18 years of age at the time of signing the Informed Consent Form (ICF) and have a life expectancy of at least 3 months.
* Karnofsky performance status of 70 or better.
* Adhere to the study visit schedule
* Voluntarily sign the Informed Consent Form (ICF).
* Baseline studies completed within 30 days of first study dose.
* Women of child-bearing potential (WCBP) defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally post-menopausal for at least 24 consecutive months must have a negative serum or urine pregnancy test within 2 weeks of first study dose and prior to each additional cycle of treatment.
* All WCBP and all sexually active male patients must agree to use adequate methods of birth control throughout the study

  ** Non-small cell lung cancer (NSCLC)enrolled in the Expansion Phase of the study must meet the following additional inclusion criteria:
* NSCLC that meets the disease criteria described in the first three Inclusion Criteria.
* Must have archival NSCLC tissue available for submission and analysis.

Exclusion Criteria:

* Treatment within 1 week of the start of IPI-504 for erlotinib, and imatinib; within 2 weeks for gefitinib, and any other tyrosine kinase inhibitor (approved or investigational); within 4 weeks for any biologic therapy (antibody, vaccine, or other protein-based therapy), radiation therapy, or conventional chemotherapy; within 6 weeks for nitrosoureas or mitomycin C.
* Radiation therapy within 2 weeks of the start of IPI-504. (Patients must have recovered from any toxicities.)
* Concurrent radiation therapy or treatment with any other investigational agent is not permitted.
* Use of a medication or food that is a clinically relevant CYP3A inhibitor or inducer within 2 weeks prior to Cycle 1, Dose 1.
* Symptomatic peripheral neuropathy ≥ Grade 2.
* Inadequate hematologic function defined by absolute neutrophil count (ANC) <1,500 cells/mm3, a platelet count <100,000/mm3, and a hemoglobin <9.0 g/dL (may be increased to this level with transfusion as long as there is no evidence of active bleeding).
* Inadequate renal function defined by AST and/or ALT >1.5; total bilirubin above the upper limit of normal.
* Inadequate renal function defined by serum creatinine >1.5 x ULN.
* Sinus bradycardia (resting heart rate <50) secondary to intrinsic conduction system disease. Patients with sinus bradycardia secondary to pharmacologic treatment may enroll if withdrawal of the treatment results in normalization of the resting heart rate to within normal limits.
* Baseline QTc >450 msec in males; QTc >470 msec in females, or previous history of QT prolongation while taking other medications.
* Presence of left bundle branch block, right bundle branch block plus left anterior hemiblock, bifasicular block or 3rd degree heart block. This does not include patients with a history of these events with adequate control by pacemaker.
* Patients who have received >450 mg/m2 of any anthracycline during prior chemotherapy must have a baseline LVEF >40%.
* Active keratitis or keratoconjunctivitis.
* History of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.
* Presence of active infection or systemic use of antibiotics within 72 hours of treatment.
* Untreated brain metastases. Note: Patients with a history of brain metastases are eligible as long as definitive treatment has been given and patients are clinically stable.
* Significant co-morbid condition or disease which in the judgment of the Investigator would place the patient at undue risk or interfere with the study (e.g., cardiac disease such as acute coronary syndrome or unstable angina within 6 months, uncontrolled hypertension, arrhythmia requiring medication or mechanical control, cirrhotic liver disease, or other conditions).
* Previous or current malignancies at other sites within the last 2 years, with exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.
* HIV-positive patients receiving combination antiretroviral therapy.
* Women who are pregnant or lactating.
* Previous treatment with 17-AAG, DMAG, or other known Hsp90 inhibitor.
* Patients with prior hepatic resection or hepatic-directed therapy (e.g., chemoembolization or Theresphere).

  **Patients with non-small cell lung cancer (NSCLC)enrolled in the Expansion Phase of the study must meet the following additional exclusion criteria:
* Prior treatment with docetaxel
* Three or more chemotherapy regimens for metastatic disease. Note: Any number of prior treatment regimens with tyrosine kinase inhibitors is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety, maximum tolerated dose(MTD)of IPI-504 in combination with docetaxel in patients with advanced solid tumors and recommend the Phase II dose of the combination of drugs. | Weekly

SECONDARY OUTCOMES:
To determine the pharmacokinetics (PK) and response rate (CR+PR) for patients with measurable lesions (as determine by RECIST) | Weekly
To determine the pharmacokinetics (PK) of IPI-504 and docetaxel | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Riely, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - TGen Clinical Research in Scottsdale, Scottsdale, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Gabrail Cancer Center, Dover, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania